CLINICAL TRIAL: NCT01838928
Title: Minimum Effective Concentration of Bupivacaine in Ultrasound-guided Axillary Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Leonardo Henrique Cunha Ferraro, M.D., Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: FU 002
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Pain
Keywords: Axillary brachial plexus block; Ultrasound; Minimum effective concentration; Bupivacaine; ultrasound-guided axillary brachial plexus block
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Investigator

ARMS (1):
- Bupivacaine (Experimental)
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine

SUMMARY:
Background: The use of ultrasound in regional anesthesia enables a reduction in the local anesthetic volume. The present study aimed to determine the minimum effective concentration (EC50 and EC95) of bupivacaine for axillary brachial plexus block (ABPB). Methods: Following approval by the Research Ethics Committee, patients with a physical condition of I or II according to the American Society of Anesthesiologists, between 21 and 65 years of age were recruited and subjected to elective surgery of the hand and ABPB. The concentration of the anesthetic was determined using a step-up/step-down method and was based on the outcome of the preceding block.

DETAILED DESCRIPTION:
The demographic data of all included patients were recorded. Routine monitoring of the surgical procedure, including electrocardiography, non-invasive blood pressure and pulse oximetry, was performed. Peripheral venous access was established in the nonoperative upper limb and standard intravenous premedication (0.03 mgkg of midazolan) was administered to all patients.

Brachial plexus blocks were performed through the axilla on patients in a supine position using a ultrasound device with a 13-6 MHz linear transducer (SonoSite, Bothell, WA, USA) and a Stimuplex® DIG RC peripheral nerve stimulator (B. Braun, Melsung, Germany).

The end of the local anesthetic injection was considered time 0 for evaluating the effectiveness of the block. A blinded observer, who was not present during the injection and was unaware of the concentration of local anesthetic used, assessed motor, thermal and sensory blocks. These assessments were performed every 5 minutes after the procedure for 30 minutes or until the block was deemed effective.

Motor function was assessed using a modified Bromage scale. The following muscles were assessed: finger flexors (median nerve), finger extensors (radial nerve), finger adductors (ulnar nerve) and elbow flexion (musculocutaneos nerve).The assessment of thermal sensation in the upper limb was performed using gauze and alcohol. Pain sensation was assessed by a pinprick test using a 23 G needle. The thermal and pain sensitivities of the ulnar, median, radial and musculocutaneos were examined.

Surgical anesthesia was defined as a motor scale of 2 or lower, with absent of appreciation of cold and pinprick sensation. Patients who exhibited block failure received an ultrasound-guided complement to the nerve block distal to axilla or conversion to general anestehesia.

All patients received a subcutaneous injection of 3 mL of a 2% lidocaine solution with epinephrine as a supplementary intercostobrachial block due to the use of a pneumatic tourniquet on the middle third of the arm. During surgery, an infusion of 25-50 mcg.kg-1.min-1 of propofol was used to achieve proper sedation.

Postoperative analgesia was assessed in the recovery room using a numeric pain rating scale (0 indicating no pain, 10 indicating the worst pain ever experienced) and the amount of analgesic used at four hours after the ABPB.

After the surgical procedure, the patients were admitted to the recovery room, where they were monitored until they met the conditions for discharge into an outpatient regimen.

Statistical Analysis

In this study, the primary objective was to estimate the minimum effective concentration of a 5-mL bupivacaine solution without epinephrine for ultrasound-guided ABPB. Volume assignment was carried out using a biased coin design up-and-down sequential method.The initial concentration of local anesthetic was 0.35%. This dose was chosen based on our clinical experience and statistical simulation at various doses. Each subsequent dose was based on the response of the preceding subject, as per a biased-coin design up-down sequential method.6 The dosing changes were in increments of 0,05%. The anesthesia provider was blinded to the concentration of bupivacaine, as was the subject. If a failure was observed in the previous subject, the dose was stepped up in the next subject. If a success was observed, the next subject was randomized with probability of 0.1 to the next lower dose and with probability of 0.9 to the same dose.

The ED95 with 95% confidence intervals (CIs) and estimated probabilities were calculated using logistic regression with SAS software. A sample size of at least 40 patients was selected after testing a variety of scenarios, each with simulations of both the responses and the corresponding doses selected by the sequential allocation method described above, and beginning with various starting doses.

The means and standard deviations were used to analyse parametric data, whereas medians and quartiles were used to analyse non-parametric data.

ELIGIBILITY:
Inclusion Criteria:

* patients with a physical condition of I or II according to the American Society of Anesthesiologists,
* between 18 and 65 years of age
* unilateral hand surgery
* BMI< 35 kg;m@

Exclusion Criteria:

* contraindication to regional anesthesia
* bleeding diathesis
* inability to visualize one or more nerves in the axilla
* psychiatric history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Minimum effective concentration of bupivacaine in ultrasound-guided axillary brachial plexus block | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo HC Ferraro, M.D., Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Takeda A, Ferraro LH, Rezende AH, Sadatsune EJ, Falcao LF, Tardelli MA. Minimum effective concentration of bupivacaine for axillary brachial plexus block guided by ultrasound. Braz J Anesthesiol. 2015 May-Jun;65(3):163-9. doi: 10.1016/j.bjane.2013.11.007. Epub 2015 Feb 16. PMID 25925026